CLINICAL TRIAL: NCT00689507
Title: A Phase 1 Safety Study of LY2127399 in Combination With Bortezomib in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Phase 1 Safety Study of LY2127399 in Combination With Bortezomib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Applied Molecular Evolution (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H9S-MC-JDCF
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed; Refractory; Bortezomib; Velcade
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — tabalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Escalation Phase(Part A): (Experimental): 1,10, 30, 100 or 300 mg of LY2127399 IV on day 1 of specific 21 day cycles and 1.3 mg/m2 Bortezomib IV on days 1, 4, 8, and 11 of each 21 day cycle
  Interventions: Biological: LY2127399
- Dose Confirmation Phase (Part B1): (Experimental): Dose determined by PK/PD modeling, LY2127399 IV on day 2 of Cycle 1 and on day 1 of specific cycles and 1.3 mg/m2 Bortezomib IV on days 1, 4, 8, and 11 of each cycle
  Interventions: Biological: LY2127399
- Dose Confirmation Phase (Part B2): (Experimental): Dose determined by PK/PD modeling, LY2127399 IV on day 1 of specific cycles and 1.3 mg/m2 Bortezomib IV on days 1, 4, 8, and 11 of specific cycles
  Interventions: Biological: LY2127399

INTERVENTIONS:
Biological: LY2127399 — monoclonal antibody

SUMMARY:
H9S-MC-JDCF was a multicenter non-randomized, single-arm, open-label, dose-escalation, dose confirmation, Phase 1 study of intravenous (IV) LY2127399 in combination with bortezomib in patients with refractory or relapsed MM.

DETAILED DESCRIPTION:
This is a study of a drug known as LY2127399, which will be given with a common treatment for multiple myeloma called bortezomib (Velcade). The primary purpose of this study is to (1)Determine the safety of LY2127399 in combination with bortezomib and any side effects that might be associated with it; (2)Assess whether LY2127399 in combination with bortezomib may help patients with relapsed or refractory multiple myeloma; (3)How much LY2127399 should be given to patients along with bortezomib.

ELIGIBILITY:
Inclusion Criteria:

* Have relapsed or refractory multiple myeloma treated with at least 1 prior regimen. Prior therapy with bortezomib is allowed if there has been no relapse or progression within 3 months of the last dose of bortezomib, and bortezomib is considered by the treating physician to be a reasonable therapy for the patient.
* Have measurable disease defined by one or more of the following:

  * Monoclonal protein in the serum of ≥1 g/dL (10 g/L).
  * Monoclonal light chain in the urine protein electrophoresis of ≥ 200 mg/24 hours.
  * Involved Serum Free Light Chain (SFLC) level > 10 mg/dL (100 mg/L) provided SFLC ratio is abnormal.
  * Measurable plasmacytoma.
* Are ≥ 18 years of age.
* Have given written informed consent prior to any study-specific procedures
* Have adequate organ function including:

  * Absolute neutrophil count (ANC) ≥ 1000/microliter
  * Platelet (PLT) count ≥ 50,000/microliter
  * Hemoglobin (Hgb) ≥ 8.0 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (if total is elevated check direct and, if normal, patient is eligible)
  * Aspartate transaminase (AST) ≤ 3 x ULN
  * Creatinine ≤ 3.0 mg/dl.
* Have a performance status of ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) scale (refer to Attachment JDCF.5).
* Have discontinued all previous therapies for cancer, including chemotherapy and radiotherapy at least 2 weeks (6 weeks for mitomycin-C or nitrosoureas) prior to study enrollment and recovered from the acute effects of therapy.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 4 months following the last dose of study drug.
* Females with child bearing potential must have had a negative urine or serum pregnancy test ≤ 3 days prior to the first dose of study drug.
* Have an estimated life expectancy of ≥ 16 weeks.
* Treatment with prior autologous transplant is permitted. If a transplant is used as consolidation following chemotherapy, without intervening disease progression, it will be considered one line of treatment with the preceding chemotherapy.

Exclusion Criteria:

* Have received treatment within 30 days of the initial dose of study drug with a drug that has not received regulatory approval for any indication.
* Have one or more serious preexisting medical conditions that, in the opinion of the investigator, would preclude participation in this study.
* Have uncontrolled infection.
* Females who are pregnant or lactating.
* Have known positive test results in human immunodeficiency virus (HIV), hepatitis B surface antigen (HBSAg), or hepatitis C antibodies (HCAb).
* Have peripheral neuropathy of > Grade 2, or of any grade with pain, as measured by CTCAE v3.0.
* Previously treated with LY2127399, or have had significant allergy to humanized monoclonal antibodies that, in the opinion of the investigator, poses an increased risk to the patient.
* Prior allogeneic hematopoietic stem cell transplant.
* Prior therapy with experimental agents targeting BAFF.
* Have QTc interval > 450 msec on baseline 12-lead ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-03; Primary Completion 2013-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK)/Pharmacodynamic (PD)modeling of LY2127399 to determine a Phase 2 dose | 2 years

SECONDARY OUTCOMES:
Safety and toxicity profile for LY2127399 in combination with bortezomib | 2 years
Response rate, duration of response, and time to progression of LY2127399 in combination with bortezomib | 2 years
Response rate, duration of response, and time to progression of LY2127399 as a single-agent | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Carpenter, PhD, Study Director — Applied Molecular Evolution
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - UCLA, Los Angeles, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania